CLINICAL TRIAL: NCT03232723
Title: Imaging Non-brain Electromagnetic Activity in Healthy Adults Using MEG
Acronym: BODMEG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 17-00684
Record Dates: First submitted 2017-07-25; First posted 2017-07-28 (Actual); Last update posted 2019-06-05 (Actual); Status verified 2019-06

CONDITIONS: Chronic Pain
Keywords: Magnetoencephalography; Whole-cortex MEG System (with optional EEG)
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- MEG Recording (Other): Magnetic fields will be recorded using a 275-channel whole-head MEG system
  Interventions: Diagnostic Test: Whole-cortex MEG System (with optional EEG)

INTERVENTIONS:
Diagnostic Test: Whole-cortex MEG System (with optional EEG) — "Whole-Cortex MEG System" non- invasively measures the magnetoencephalographic (MEG) signals (and, optionally, electroencephalographic EEG signals) produced by electrically active tissue of the brain. These signals are recorded by a computerized data acquisition system, displayed, and may then be interpreted by trained physicians to help localize these active areas. The location may then be correlated with anatomical information of the brain. MEG is routinely used to identify the locations of visual, auditory, somatosensory, and motor cortex in the brain.

SUMMARY:
The primary purpose of this study is to determine the effectiveness of the Magnetoencephalography (MEG) instrument to record electrical activity from parts of the body other than the brain. This study will examine if electrical activity from parts of the body, other than the brain, can be imaged by the MEG instrument. Finding will contribute to studies of pain, since abnormal electrical activity in skeletal muscle is the basis of pain, which can be severe, yet there is no non-invasive way to image this abnormal activity. This is particularly relevant to deep muscle pain and back pain.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults who are willing and able to provide informed consent.

Exclusion Criteria:

* Subjects with characteristics incompatible with MEG recordings as listed on the MEG Safety checklist (Appendix A),
* Involuntary, uncontrolled tremor,
* chronic pain.
* pregnant women (based on self-report).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2017-09-07 (Actual); Study Completion 2017-09-07 (Actual)

PRIMARY OUTCOMES:
Determination of optimal position to obtain safe and effective imaging of structures other than the brain. | 2 Weeks
  * Hand position 1 relaxed
  * Hand position 1 muscles active
  * Hand position 2 relaxed
  * Hand position 2 muscles active
  * Neck and Jaw, relaxed
  * Neck and Jaw, tensed
  * Upper torso relaxed
  * Area of interest 1 relaxed(areas are not specific for Runs 9-11. (Possible areas are groups of muscles in the back and limbs.)
  * Area of interest 1 tensed(areas are not specific for Runs 9-11. (Possible areas are groups of muscles in the back and limbs.)
  * Area of interest 2 relaxed(areas are not specific for Runs 9-11. (Possible areas are groups of muscles in the back and limbs.)
  * Area of interest 2 tensed (areas are not specific for Runs 9-11. (Possible areas are groups of muscles in the back and limbs.)
Evoked activity to obtain safe and effective imaging of structures other than the brain | 2 Weeks
  * Hand position 1 relaxed
  * Hand position 1 muscles active
  * Hand position 2 relaxed
  * Hand position 2 muscles active
  * Neck and Jaw, relaxed
  * Neck and Jaw, tensed
  * Upper torso relaxed
  * Area of interest 1 relaxed(areas are not specific for Runs 9-11. (Possible areas are groups of muscles in the back and limbs.)
  * Area of interest 1 tensed(areas are not specific for Runs 9-11. (Possible areas are groups of muscles in the back and limbs.)
  * Area of interest 2 relaxed(areas are not specific for Runs 9-11. (Possible areas are groups of muscles in the back and limbs.)
  * Area of interest 2 tensed (areas are not specific for Runs 9-11. (Possible areas are groups of muscles in the back and limbs.)

SECONDARY OUTCOMES:
Dominant frequency of non-brain electrical activity in healthy adults. | 2 Weeks
  * Hand position 1 relaxed
  * Hand position 1 muscles active
  * Hand position 2 relaxed
  * Hand position 2 muscles active
  * Neck and Jaw, relaxed
  * Neck and Jaw, tensed
  * Upper torso relaxed
  * Area of interest 1 relaxed(areas are not specific for Runs 9-11. (Possible areas are groups of muscles in the back and limbs.)
  * Area of interest 1 tensed(areas are not specific for Runs 9-11. (Possible areas are groups of muscles in the back and limbs.)
  * Area of interest 2 relaxed(areas are not specific for Runs 9-11. (Possible areas are groups of muscles in the back and limbs.)
  * Area of interest 2 tensed (areas are not specific for Runs 9-11. (Possible areas are groups of muscles in the back and limbs.)
Location of non-brain of activity in healthy adults. | 2 Weeks
  * Hand position 1 relaxed
  * Hand position 1 muscles active
  * Hand position 2 relaxed
  * Hand position 2 muscles active
  * Neck and Jaw, relaxed
  * Neck and Jaw, tensed
  * Upper torso relaxed
  * Area of interest 1 relaxed(areas are not specific for Runs 9-11. (Possible areas are groups of muscles in the back and limbs.)
  * Area of interest 1 tensed(areas are not specific for Runs 9-11. (Possible areas are groups of muscles in the back and limbs.)
  * Area of interest 2 relaxed(areas are not specific for Runs 9-11. (Possible areas are groups of muscles in the back and limbs.)
  * Area of interest 2 tensed (areas are not specific for Runs 9-11. (Possible areas are groups of muscles in the back and limbs.)

CONTACTS AND LOCATIONS:
Overall Officials: Rodolfo Llinas, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided